CLINICAL TRIAL: NCT01576783
Title: Omega Tots: A Randomized, Controlled Trial of Long-chain Polyunsaturated Fatty Acid Supplementation of Toddler Diets and Developmental Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sarah Keim (Other)
Collaborators: Allen Foundation Inc. (Other); March of Dimes (Other); Cures Within Reach (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Sarah Keim, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 183210
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Preterm Birth; Child Development
MeSH Terms: conditions — Premature Birth | interventions — Docosahexaenoic Acids; Arachidonic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docosahexaenoic Acid + Arachidonic Acid (Experimental): Docosahexaenoic Acid + Arachidonic Acid (DHA+AA)
  Interventions: Drug: Docosahexaenoic Acid + Arachidonic Acid (DHA+AA)
- Placebo (Placebo Comparator): Corn oil supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Docosahexaenoic Acid + Arachidonic Acid (DHA+AA) — 200 mg DHA+ 200 mg AA per day for 6 months
  Arms: Docosahexaenoic Acid + Arachidonic Acid
Dietary Supplement: Placebo — 400 mg corn oil per day for 6 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether supplementation with certain polyunsaturated fatty acids can help the cognitive development of children born preterm.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-16 completed months (age corrected for prematurity) at baseline
2. Discontinued regular breastfeeding and formula feeding at the time of randomization
3. Gestational age < 35 completed weeks at birth
4. English is primary language in home
5. Informed consent obtained and signed
6. Child admitted to any NCH managed NICU or children who have ever had a Neonatology Clinic follow up visit scheduled, regardless of attendance

Exclusion Criteria:

1. Feeding problems
2. Major malformation, metabolic, or digestive disorder that would preclude participation and/or optimal absorption of the supplement.
3. Weight < 5th or > 95th percentile for age, per WHO growth charts
4. Consume DHA supplement drops, chews, or powders or Pediasure, or fatty fish more than 2x per week
5. Plans to move out of the area within the next 6 months
6. Known corn allergy
7. Known soy allergy
8. Known fish allergy

Ages: 10 Months to 16 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 377 (Actual)
Dates: Start 2012-04-26 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Keim, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Boone KM, Pattison K, Pelak G, Sheppard KW, Rausch J, Yeates KO, Nelin MA, Klebanoff MA, Turner AN, Rogers LK, Keim SA. Docosahexaenoic and arachidonic acid supplementation at 1 year has mixed effects on development and behaviour at age 2 for preterm children. Acta Paediatr. 2021 Jul;110(7):2082-2083. doi: 10.1111/apa.15858. Epub 2021 Apr 12. No abstract available. PMID 33768637
- [Derived] Sullivan JA, Wiese AM, Boone KM, Rausch J, Keim SA. To attend, or not to attend: Examining caregiver intentions and study compliance in a pediatric, randomized controlled trial. Clin Trials. 2020 Apr;17(2):223-230. doi: 10.1177/1740774519893307. Epub 2020 Jan 27. PMID 31984781
- [Derived] Boone KM, Rausch J, Pelak G, Li R, Turner AN, Klebanoff MA, Keim SA. Docosahexaenoic Acid and Arachidonic Acid Supplementation and Sleep in Toddlers Born Preterm: Secondary Analysis of a Randomized Clinical Trial. J Clin Sleep Med. 2019 Sep 15;15(9):1197-1208. doi: 10.5664/jcsm.7902. PMID 31538590
- [Derived] Boone KM, Nelin MA, Chisolm DJ, Keim SA. Gaps and Factors Related to Receipt of Care within a Medical Home for Toddlers Born Preterm. J Pediatr. 2019 Apr;207:161-168.e1. doi: 10.1016/j.jpeds.2018.10.065. Epub 2018 Dec 19. PMID 30579584
- [Derived] Keim SA, Boone KM, Klebanoff MA, Turner AN, Rausch J, Nelin MA, Rogers LK, Yeates KO, Nelin L, Sheppard KW. Effect of Docosahexaenoic Acid Supplementation vs Placebo on Developmental Outcomes of Toddlers Born Preterm: A Randomized Clinical Trial. JAMA Pediatr. 2018 Dec 1;172(12):1126-1134. doi: 10.1001/jamapediatrics.2018.3082. PMID 30357263

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Started | 189 | 188
Completed | 169 | 171
Not Completed | 20 | 17
Not completed — Change in Medical Care | 1 | 0
Not completed — Lost to Follow-up | 14 | 16
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo | Total
Number analyzed (Participants) | 189 | 188 | 377
Age, Continuous [Median (Inter-Quartile Range); unit: Months] — Maximum age was 16 completed months, meaning someone who was 16 months and 29 days could be eligible to participate because they did not reach 17 months
  Months | 15.7 [13.8 to 16.5] | 15.6 [13.1 to 16.5] | 15.7 [13.6 to 16.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 98 | 182
  Male | 105 | 90 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 17
  Not Hispanic or Latino | 182 | 178 | 360
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 52 | 53 | 105
  White | 114 | 122 | 236
  More than one race | 21 | 12 | 33
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 189 | 188 | 377

OUTCOME MEASURES:

1. Primary Outcome: Erythrocyte Fatty Acid Levels
Description: This outcome measure involved an examination of change in plasma and RBC fatty acid concentrations from the first study visit to the final study visit. The changes were calculated as the fatty acid level at 180 days minus the fatty acid level at baseline. Primary Outcome for 1st stage of project funded by Allen Foundation, Inc
Time Frame: Baseline to 180 days post-randomization
Population: Rows titles are fatty acids with different C:D ratio where, "C"= Carbohydrate; "D" = Double bond; "C:D" is the ratio of the total amount of Carbon atoms of the fatty acid in relation to the number of double (unsaturated) bonds in it. Funding allotted for 205 children to be randomized to provide blood specimens but only 173 gave pre and post samples
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 85 | 88
nmol/mL
  Linoleic acid (18:2n-6) | -2.1 (5.2) | 0.6 (4.4)
  Arachidonic acid (20:4n-6) | 2.0 (2.6) | -0.2 (1.1)
  Total n-6 | 0.2 (6.0) | 0.4 (5.0)
  α-linolenic acid (18:3n-3) | -0.1 (0.4) | 0.0 (0.3)
  Eicosapentaenoic acid (20:5n-3) | 0.0 (0.1) | -0.1 (0.2)
  Docosapentaenoic acid (22:5n-3) | -0.1 (0.1) | 0.0 (0.1)
  Docosahexaenoic acid (22:6n-3) | 1.1 (1.0) | -0.1 (0.2)
  Total n-3 | 0.9 (1.1) | -0.2 (0.5)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; The change in erythrocyte fatty acids and the change in dietary DHA and EPA (aside from the supplement) were examined by treatment group using mixed effects regression, again with a random-effect for within-family dependence; Test type: Other — The reported p-value is for the comparison of the change in Linoleic acid (18:2n-6) mol% between groups (DHA+AA vs. Placebo); p < 0.001, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.4 to 0.9]
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in Arachidonic acid (20:4n-6) mol% between groups (DHA+AA vs. Placebo); p < 0.001, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = 2.2, 95% CI 2-sided [1.7 to 2.8]
Statistical Analysis 3: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in Total n-6 mol% between groups (DHA+AA vs. Placebo); p = 0.61, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.0 to 1.7]
Statistical Analysis 4: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in α-linolenic acid (18:3n-3) between groups (DHA+AA vs. Placebo); p = 0.40, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 5: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in Eicosapentaenoic acid (20:5n-3) between groups (DHA+AA vs. Placebo); p = 0.12, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.1]
Statistical Analysis 6: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in Docosapentaenoic acid (22:5n-3) between groups (DHA+AA vs. Placebo); p < 0.001, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.1 to 0.0]
Statistical Analysis 7: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in Docosahexaenoic acid (22:6n-3) between groups (DHA+AA vs. Placebo); p < 0.001, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = 1.2, 95% CI 2-sided [1.0 to 1.5]
Statistical Analysis 8: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in Total n-3 between groups (DHA+AA vs. Placebo); p < 0.001, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.9 to 1.4]

2. Primary Outcome: Erythrocyte Fatty Acid Levels (Additional Data)
Description: as for outcome 1
Time Frame: Baseline to 180 days post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 85 | 88
ratio | -3.2 (3.9) | 1.6 (2.8)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in n-6:n-3 ratio between groups (DHA+AA vs. Placebo); p < 0.001, Mixed Models Analysis — Threshold for statistical significance (<0.05); Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-5.5 to -3.7]

3. Primary Outcome: Enrollment and Trial Completion
Description: The number of children who enroll in the trial and the number of those children who return for study visits 2 and 3. Primary Outcome for 1st stage of project funded by Allen Foundation, Inc.
Time Frame: Baseline to 180 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 189 | 188
Participants
  Study Visit 2 Completion | 172 | 163
  Study Visit 3 Completion | 166 | 168

4. Primary Outcome: Adherence
Description: The mean (average) percentage of packets consumed by the children assigned to the supplement or placebo. Primary Outcome for 1st stage of project funded by Allen Foundation, Inc
Time Frame: Baseline to 180 days post-randomization
Measure: Mean (Standard Deviation); unit: average percentage of packets consumed
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 189 | 188
average percentage of packets consumed | 80.6 (28) | 80.7 (25)

5. Secondary Outcome: (Behavior) Infant Behavior Questionnaire-Revised (IBQ-R; Short Form)
Description: Infant Behavior Questionnaire-Revised (IBQ-R; short form) was used to assess effortful control (12 items) and activity level (3 items). The IBQ-R measures early temperament-based inhibitory control,a key component of executive function as children mature. Scores range from 1 to 7, with higher scores indicating greater frequency of behaviors. IBQ-R scores were measured at baseline and then again at study completion (180 days post randomization). The scores were calculated as a change between two time points (the IBQ-R value at 180 days minus the IBQ-R value at baseline).
Time Frame: Baseline to 180 days post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 189 | 188
units on a scale
  Effortful Control | -0.7 (0.8) | -0.5 (0.8)
  Activity Level | 0.6 (1.5) | 0.5 (1.5)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in Effortful Control Composite scores between groups (DHA+AA vs. Placebo); p = .13, Mixed Models Analysis — Threshold for statistical significance (<0.05); Analyses compared the change in scores between groups, using mixed effects regression that leveraged maximum likelihood to include missing data
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in Activity Level Composite scores between groups (DHA+AA vs. Placebo); p = .76, Mixed Models Analysis — Threshold for statistical significance (<0.05)

6. Secondary Outcome: (Development) Bayley Scales of Infant and Toddler Development, Third Edition(Bayley-III)
Description: Bayley Scales of Infant and Toddler Development, third edition, (Bayley-III) is an instrument designed to measure the developmental functioning of infants and toddlers between the ages of 1 month and 42 months (age adjustments for prematurity are accommodated with the tool). It provides age specific composite scores for cognitive (91 items,score min 55 max 145), language (98 items, score min 47 max 153), and motor (138 items, score min 46 max 154) skills. For all scales, higher scores are better and lower scores indicate possible delay/deficit. Bayley-III scores were measured at baseline and then again at study completion (180 days post randomization). The scores were calculated as a change between two time points (the Bayley-III value at 180 days minus the Bayley-III value at baseline). Secondary Outcome for 1st stage of project funded by Allen Foundation, Inc; Primary Outcome for 2nd stage of project funded by March of Dimes and Health Resources and Services Administration
Time Frame: Baseline to 180 days post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 189 | 188
units on a scale
  Cognitive Composite | -2.6 (13.3) | -3.7 (12.2)
  Language Composite | -0.5 (12.0) | 0.2 (12.6)
  Motor Composite | -0.6 (12.5) | -0.4 (12.7)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; A sample of 448 was planned to achieve >80% power to detect a 4.2-point difference (0.27-standard deviation (SD)) in Bayley-III cognitive composite scores with 10% loss to follow-up.The investigational product manufacturer discontinued production once 377 were enrolled, thereby capping enrollment. That sample provided 80% power to detect a 0.29-SD difference in Bayley-III scores; Test type: Other — The reported p-value is for the comparison of the change in Cognitive Composite scores between groups (DHA+AA vs. Placebo); p = .66, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in Language Composite scores between groups (DHA+AA vs. Placebo); p = .55, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Other — The reported p-value is for the comparison of the change in Motor Composite scores between groups (DHA+AA vs. Placebo); p = .88, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 5, analysis 1]

7. Other Pre Specified Outcome: Brief Infant Sleep Questionnaire (BISQ)
Description: The following sleep characteristics were captured based on caregiver-report: nocturnal sleep duration (hours), daytime sleep duration (hours), total sleep duration within a 24-hour period (hours). Larger values represent more time spent in each type of sleep. BISQ scores were measured at baseline and then again at study completion (180 days post randomization). The scores were calculated as a change between two time points (the BISQ value at 180 days minus the BISQ value at baseline).
Time Frame: Baseline to 180 days post-randomization
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 189 | 188
hours
  Nocturnal Sleep Duration | 0.25 (1.61) | -0.16 (1.34)
  Daytime Sleep Duration | -0.32 (1.15) | -0.46 (1.25)
  Total Sleep Duration | -0.07 (2.22) | -0.57 (1.7)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in Nocturnal Sleep Duration between groups (DHA+AA vs. Placebo); p = .11, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in daytime sleep duration between groups (DHA+AA vs. Placebo); p = 0.47, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in total sleep duration between groups (DHA+AA vs. Placebo); p = 0.32, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 5, analysis 1]

8. Other Pre Specified Outcome: Body Composition
Description: Changes in body composition from baseline to 6 months post-randomization (weight, recumbent length, head circumference, mid-upper arm circumference, triceps and subscapular skinfolds). These measurements were converted to z scores for corrected age based on Child Growth Standards from the World Health Organization. The z-score indicates the number of standard deviations away from the mean. A z score of 0 is equal to the mean of a reference population (children the same age and sex). Values less than 0 indicate values lower than the reference population, while values greater than 0 indicate values higher than the reference population.
Time Frame: Baseline to 180 days post-randomization
Measure: Mean (Standard Deviation); unit: z scores
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 189 | 188
z scores
  Weight | 0.1 (0.4) | 0.0 (0.4)
  Recumbent Length | 0.1 (0.9) | 0.2 (0.9)
  Head Circumference | -0.0 (0.6) | -0.1 (0.5)
  Mid-Upper Arm Circumference | 0.0 (0.8) | 0.1 (0.7)
  Triceps Skinfold | -0.0 (0.7) | -0.1 (0.8)
  Subscapular Skinfold | -0.2 (0.8) | -0.2 (0.9)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in weight-for-age z scores between groups (DHA+AA vs. Placebo); p = 0.99, Mixed Models Analysis — Threshold for statistical significance (<0.05); Analyses compared the change in scores between groups, using mixed-effects regression that leveraged maximum likelihood to account for missing data
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in length-for-age z scores between groups (DHA+AA vs. Placebo); p = 0.27, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in head circumference-for-age z scores between groups (DHA+AA vs. Placebo); p = 0.39, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in mid upper arm circumference-for-age z scores between groups (DHA+AA vs. Placebo); p = 0.25, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in triceps skinfold-for-age z scores between groups (DHA+AA vs. Placebo); p = 0.85, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in subscapular skinfold-for-age z scores between groups (DHA+AA vs. Placebo); p = 0.82, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 8, analysis 1]

9. Other Pre Specified Outcome: Brief Infant Toddler Social Emotional Assessment (BITSEA)
Description: BITSEA measures socioemotional development in toddlerhood. Scores were summed to provide competence (range: 0-22) and problem (range: 0-62) scores, respectively. The problem scale is further divided into subscales: externalizing (6 items; range: 0-12), internalizing (8 items; range: 0-16), and dysregulation (8 items; range: 0-16). Additionally, 14 items comprise a red flag scale (range: 0-28). Eight items from the competence and nine items from the problem subscales are indicative of behaviors often seen in children with ASD. Each of the 17 ASD items was dichotomized to illustrate the presence (1) (i.e., competence items absent, problem items present) or absence (0) (i.e., competence items present, problem items absent) of each ASD behavior. Items were then summed to derive an ASD score (range: 0-17). Higher competence scores represent better functioning, whereas higher problem (including the problem subscales), red flag, and ASD scores were indicative of poorer functioning.
Time Frame: 180 days post-randomization
Population: The number analyzed for the competence and ASD scales differs from the overall number analyzed due to missing data on these two scales.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 161 | 153
units on a scale
  Competence: number analyzed (Participants) | 161 | 152
  Competence | 16.50 (3.09) | 16.73 (2.94)
  Problem | 9.81 (6.01) | 10.18 (6.84)
  Externalizing | 2.29 (2.06) | 2.30 (1.98)
  Internalizing | 2.04 (1.58) | 2.31 (2.10)
  Dysregulation | 3.25 (2.57) | 3.29 (2.59)
  Red Flag | 2.93 (2.48) | 3.12 (2.85)
  ASD | 4.11 (2.29) | 4.36 (2.98)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at the end of the trial; p = 0.42, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at the end of the trial; p = 0.68, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model
Statistical Analysis 3: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at the end of the trial; p = 0.78, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model
Statistical Analysis 4: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at the end of the trial; p = 0.32, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model
Statistical Analysis 5: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at the end of the trial; p = 0.97, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model
Statistical Analysis 6: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at the end of the trial; p = 0.62, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model
Statistical Analysis 7: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at the end of the trial; p = 0.69, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model

10. Other Pre Specified Outcome: Pervasive Developmental Disorders Screening Test - II, Stage 2 (PDDST-II)
Description: The PDDST-II is a clinically derived, caregiver-completed screener to assist in differentiating an ASD diagnosis from other disorders in children with developmental concerns, including those born preterm. The PDDST-II comprised 14 yes/no items that indicate the presence (1) or absence (0) of developmental concerns. Items were summed (possible range: 0-14) and higher scores represented greater developmental concern.
Time Frame: 180 days post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 160 | 153
units on a scale | 2.91 (2.35) | 3.37 (3.02)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at the end of the trial; p = 0.22, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model

11. Other Pre Specified Outcome: Other Long-term Outcomes: Sleep (BISQ)
Description: Long-term (26-32 months of age) outcomes. This will be evaluated using scores on the Brief Infant Sleep Questionnaire (BISQ).The following sleep characteristics were captured based on caregiver-report: nocturnal sleep duration (hours), daytime sleep duration (hours), total sleep duration within a 24-hour period (hours). Larger values represent more time spent in each type of sleep. BISQ scores were measured at baseline and then again at post-intervention follow-up (approximately 8 months after the trial ended). The scores were calculated as a change between two time points (the BISQ value at post-intervention follow-up minus the BISQ value at baseline).
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 136 | 125
hours
  Nocturnal Sleep Duration | -0.11 (1.68) | -0.38 (1.43)
  Daytime Sleep Duration | -0.46 (1.30) | -0.81 (1.41)
  Total Sleep Duration | -0.57 (2.20) | -1.17 (1.85)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.23, Mixed Models Analysis — Threshold for statistical significance (<0.05)
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in Daytime Sleep Duration between groups (DHA+AA vs. Placebo); p = 0.07, Mixed Models Analysis — Threshold for statistical significance (<0.05)
Statistical Analysis 3: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the change in Total Sleep Duration between groups (DHA+AA vs. Placebo); p = 0.06, Mixed Models Analysis — Threshold for statistical significance (<0.05)

12. Other Pre Specified Outcome: Other Long-term Outcomes: Sleep (CSHQ)
Description: Long-term (26-32 months of age) outcomes. This will be evaluated using the total score on a subset of 13 items from the Children's Sleep Habits Questionnaire (CSHQ). The range in total score is 13-39. A higher score is indicative of more sleep problems.
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 134 | 122
units on a scale | 18.82 (4.96) | 19.57 (5.40)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — The reported p-value is for the comparison of the scores between groups (DHA+AA vs. Placebo) at post-intervention follow-up (median of 8.3 months (IQR = 4.8) after trial completion and supplementation stopped); p = 0.51, Mixed Models Analysis — Threshold for statistical significance (<0.05); Continuous scores at the end of the trial were compared using a linear mixed model

13. Other Pre Specified Outcome: Long-term Efficacy in Improving Cognition
Description: Long-term (26-32 months of age) cognitive outcome. This will be evaluated based on standard scores from the cognitive section of the Developmental Profile - 3. The range in standard scores is 40-140 with higher scores represent better cognitive ability.
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 134 | 120
units on a scale | 103.36 (19.00) | 107.93 (19.93)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.09, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups. Model controlled for baseline scores

14. Other Pre Specified Outcome: Long-term Efficacy in Improving Executive Functions (BRIEF-P)
Description: Long-term (26-32 months of age) executive function outcomes. This will be evaluated using scores on the Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P). The BRIEF-P yields five clinical scales, each measuring a different aspect of executive function: inhibit, shift, emotional control, working memory, and plan/organize. The clinical scales merge to create four broad indices of executive function: inhibitory self-control, flexibility, emergent metacognition, and global executive composite. A t-score of 50 is equal to the population mean with scores below 50 indicating better executive function, and scores above 50 indicating worse executive function for each reported aspect.
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 115 | 104
units on a scale
  Inhibit | 50.20 (10.69) | 51.91 (10.57)
  Shift | 47.08 (8.89) | 49.16 (9.92)
  Emotional Control | 48.55 (8.20) | 49.98 (9.33)
  Working Memory | 53.79 (11.30) | 56.04 (13.63)
  Plan/Organize | 49.66 (10.58) | 52.69 (12.02)
  Inhibitory Self-control Index | 49.44 (9.44) | 51.13 (10.23)
  Flexibility Index | 47.62 (8.72) | 49.60 (9.88)
  Emergent Metacognition Index | 52.17 (11.27) | 55.01 (13.76)
  Global Executive Composite | 50.09 (10.60) | 52.67 (12.51)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.29, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.11, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.23, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups
Statistical Analysis 4: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.29, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups
Statistical Analysis 5: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.06, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups
Statistical Analysis 6: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.14, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups
Statistical Analysis 7: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.13, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups
Statistical Analysis 8: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.16, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups

15. Other Pre Specified Outcome: Long-term Efficacy in Improving Executive Functions (CBCL)
Description: Long-term (26-32 months of age) executive function outcomes. This will be evaluated using scores on the Attention Deficit/Hyperactivity Problems DSM oriented subscale and the Attention syndrome subscale of the Child Behavior Checklist 1.5-5 (CBCL). A t-score of 50 is equal to the population mean with scores below 50 indicating less behavioral problems, and scores above 50 indicating more behavioral problems.
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 136 | 125
t-score
  Attention Deficit/Hyperactivity Problems | 55.04 (6.90) | 55.08 (6.43)
  Attention Problems | 55.21 (7.10) | 55.71 (6.82)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.98, Mixed Models Analysis; Linear mixed models compared continuous scores at follow-up between treatment groups
Statistical Analysis 2: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.67, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups

16. Other Pre Specified Outcome: Other Long-term Outcomes: Pervasive Developmental Problems
Description: Long-term (26-32 months of age) outcomes. This will be evaluated using scores on the Pervasive Developmental Problems DSM oriented scale on the Child Behavior Checklist 1.5-5 (CBCL). A t-score of 50 is equal to the population mean with scores below 50 indicating less problems and scores above 50 indicating more problems.
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 136 | 125
t-score | 53.76 (6.12) | 55.54 (7.78)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.047, Mixed Models Analysis — Threshold for statistical significance (<0.05); Linear mixed models compared continuous scores at follow-up between treatment groups

17. Other Pre Specified Outcome: Other Long-term Outcomes: Language
Description: Long-term (26-32 months of age) outcomes. This will be evaluated using scores on the Communicative Development Inventory (CDI). On this measure, caregivers selected the number of words from a list of 100 common words that their child used. Scores reflect the total number of words, from the list of 100, that the child used.
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 136 | 124
words | 56.68 (28.75) | 61.15 (27.94)
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.20, Mixed Models Analysis — Threshold for statistical significance (<0.05); [statistical method as in outcome 13, analysis 1]

18. Other Pre Specified Outcome: Other Long-term Outcomes: Number of Participants With Developmental Delay
Description: Long-term (26-32 months of age) outcomes. This will be evaluated using caregiver reports/diagnoses of developmental delay.
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Count of Participants; unit: Participants
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 133 | 116
Participants | 30 | 18
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — Results are the comparison of proportion of those with a developmental condition between groups (DHA+AA vs. Placebo) at post-intervention follow-up (median of 8.3 months (IQR = 4.8) after trial completion and supplementation stopped); Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.80 to 3.32]

19. Other Pre Specified Outcome: Other Long-term Outcomes: Number of Participants With Behavior Difficulties
Description: Long-term (26-32 months of age) outcomes. This will be evaluated using caregiver reports/diagnoses of behavioral difficulties.
Time Frame: Long-term effect (approximately 8 months) after intervention completion
Measure: Count of Participants; unit: Participants
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
Number analyzed (Participants) | 133 | 116
Participants | 5 | 1
Statistical Analysis 1: Comparison: Docosahexaenoic Acid + Arachidonic Acid vs Placebo; Test type: Other — Results are the comparison of proportion of those with a behavioral condition between groups (DHA+AA vs. Placebo) at post-intervention follow-up (median of 8.3 months (IQR = 4.8) after trial completion and supplementation stopped); Odds Ratio (OR) = 4.50, 95% CI 2-sided [0.52 to 39.15]

ADVERSE EVENTS:
Time Frame: Baseline to 180 days post randomization
Description: Information to be collected includes event description, time of onset, Study Doctor's assessment of severity, relationship to study product,and time of resolution/stabilization of the event. All AEs occurring during study participation must be documented appropriately regardless of relationship. Adverse Events were monitored/assessed and classified by body or organ system.
Arm/Group | Docosahexaenoic Acid + Arachidonic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/189 | 0/188
Serious Adverse Events (participants affected / at risk) | 0/189 | 0/188
Other Adverse Events (participants affected / at risk) | 127/189 | 129/188
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docosahexaenoic Acid + Arachidonic Acid (N=189) | Placebo (N=188)
ENT Symptoms (Ear and labyrinth disorders) | 29 | 33
Gastrointestinal Symptoms (Gastrointestinal disorders) | 69 | 63
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 23 | 22
Skin/Limb Symptoms (Skin and subcutaneous tissue disorders) | 12 | 18
Behavioral Symptoms (Social circumstances) | 22 | 19 — Includes fussiness, temper tantrums, moodiness, etc.
Misc Symptoms (Immune system disorders) | 35 | 41 — Multi-symptom illnesses reported by caregivers which typically included more than 1 body system

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT01576783/Prot_SAP_001.pdf